CLINICAL TRIAL: NCT03605394
Title: Assessment of Maxillary Sinus Septum and Its Prevalence in a Sample of Egyptian Population Using 3D CBCT : A Cross-Sectional Study
Brief Title: Assessment of Maxillary Sinus Septum and Its Prevalence in a Sample of Egyptian Population (CBCT)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farid Medhat, Assistant Professor of Oral and Maxillofacial Radiology Faculty Of Dentistry, Cairo University
Other Study IDs: RAD1:6:2
Record Dates: First submitted 2018-07-22; First posted 2018-07-30 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Maxillary Sinus
Keywords: Maxillary sinus; sinus septa; sinus septum; CBCT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
a cross-sectional study to estimate the prevalence of maxillary sinus septum and assessment of it in a sample of Egyptian Population using cone beam computed tomography through retrospective data analysis

DETAILED DESCRIPTION:
Setting and location:

1. The data collection will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University, Cairo, Egypt.
2. CBCT images will be obtained from Egyptian patients who had CBCT examination as part of their dental examination, diagnosis or treatment planning.

Participants:

A total sample of 111examined sinus belonging to Egyptian individuals will be included.

Variables:

1. Prevalence of maxillary sinus septa.
2. Location of maxillary sinus septa.
3. Orientation of maxillary sinus septa in dentulous & edentulous individual.

Data Sources / Measurements:

* Retrospective Data collection will be performed after the CBCT images are pooled from the computer database.
* All the CBCT examinations will be scanned using CBCT machine (Planmeca promax 3D Mid).
* CBCT scans using different fields of view, and different voxel resolutions .
* CBCT images will be interpreted by two oral radiologists independently; blinded from demographic data of the patients and from the results of each other.
* Each one will evaluate the images separately twice with a period of two weeks between the two reading sessions.
* Then inter-observational and intra-observational variability between the observers will be evaluated.

Bias:

No source of bias.

Study Size:

The results showed that a total sample size of 111examined sinus will be adequate to detect sinus septum prevalence of 24.6% with an 8% margin of error, a significance level of 5% and a 95% confidence interval.

Quantitative Variables:

The number of CBCT scans of Egyptian individuals with maxillary sinus septa will be counted to estimate the variations in the Egyptian population.

Statistical methods:

Data will be analysed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages.

ELIGIBILITY:
Inclusion Criteria:

* • CBCT scans of partially, fully edentulous and dentulous population.

Exclusion Criteria:

* • CBCT scans that not displaying all the extension of the lower one third of the maxillary sinus.

  * Presence of large pathological lesions involving the maxillary sinus or affecting the confines of the sinus floor.
  * Images exhibiting changes in the morphology of sinus walls due to trauma.
  * Presence of technical artifacts that make difficult the maxillary sinus evaluation.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian Population
Sampling Method: Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
prevalence of maxillary sinus septa | in the years 2017-2018-2019
  Measuring device is CBCT Software on Planmeca Promax 3D Mid,Measuring unit is Percentage

SECONDARY OUTCOMES:
Location of maxillary sinus septa | in the years 2017-2018-2019
  Measuring device is CBCT Software on Planmeca Promax 3D Mid,Measuring unit is Percentage

OTHER OUTCOMES:
Orientation of maxillary sinus septa | in the years 2017-2018-2019
  Measuring device is CBCT Software on Planmeca Promax 3D Mid,Measuring unit is Categorical data:
  * Transverse
  * Oblique
  * sagittal

IPD SHARING:
Plan to Share IPD: No